CLINICAL TRIAL: NCT06579144
Title: An Open-label, Multicentre Study to Compare the Pharmacokinetics of Efanesoctocog Alfa Versus rFVIII Products, Damactocog Alfa Pegol or Turoctocog Alfa Pegol, After a Single Intravenous Dose of 50 IU/kg in a Fixed Sequence in Previously Treated Adults With Severe Haemophilia A.
Brief Title: Pharmacokinetic Comparison of Efanesoctocog Alfa vs Other EHL-rFVIII Products in Participants With Severe Haemophilia A
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: PSI CRO (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: Sobi.BIVV001-003
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hemophilia A
Keywords: Haemophilia A; Blood coagulation disorder; efanesoctocog alfa; FVIII; Coagulation protein disorder; Pharmacokinetics
MeSH Terms: conditions — Hemophilia A; Blood Coagulation Disorders; Coagulation Protein Disorders | interventions — BIVV001

STUDY DESIGN:
Intervention Model Description: Open-label, 2-period, fixed-sequence study for intra-participant comparison of PK-profiles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Damactocog alfa pegol (Active Comparator): Patients treated with damactocog alfa pegol at the time of screening will receive one single injection with 50 IU/kg at visit 1, then one single dose 50 IU/kg with efanesoctocog alfa at visit 8.
  Interventions: Drug: Efanesoctocog alfa
- Turoctocog alfa pegol (Active Comparator): Patients treated with turoctocog alfa pegol at the time of screening will receive one single injection with 50 IU/kg at visit 1, then one single dose 50 IU/kg with efanesoctocog alfa at visit 8.
  Interventions: Drug: Efanesoctocog alfa

INTERVENTIONS:
Drug: Efanesoctocog alfa — Recombinant coagulation factor VIII Fc-von Willebrand Factor-XTEN fusion protein (rFVIIIFc-VWF-XTEN)
  Other Names: BIVV001; Altuvoct; Altuviiio

SUMMARY:
Sobi.BIVV001-003 is an open-label, 2-period, fixed sequence study for intra-participant comparison of the PK profiles of efanesoctocog alfa and the extended half-life rFVIII products damactocog alfa pegol or turoctocog alfa pegol after a single i.v. injection in previously treated males, 18-65 years of age, with severe haemophilia A.

Participants who are receiving treatment with damoctocog alfa pegol (n~12) or turoctocog alfa pegol (n~12) will be enrolled in the study. The study will start with a screening period (up to 28 days), including a wash-out period prior to start of the actual study period.

During the the first visit, a single dose of damactocog alfa pegol or turoctocog alfa pegol (corresponding to the participant's pre-study treatment) will be administered. A PK sampling period will follow over 7 visits. Following completion of the PK sampling of the original treatment regimen, the patients will be given a single dose of efanesoctocog alfa at visit 8, after which a new PK sampling period will follow (visit 8-15).

The primary objective for the study is to compare the half-life of efanesoctocog alfa with that of the two comparator drugs after a single iv. injections.

Secondary objectives include comparison of area under the curve for efanesoctocog alfa vs. the two comparator drugs, characterization of PK parameters for all three drugs as well as well as to evaluate safety and tolerability of a single iv. injection of efanesoctocog alfa.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be male, 18 to 65 years of age, inclusive, at the time of signing the informed consent form (ICF).
* Severe haemophilia A, defined as <1 IU/dL (<1%) endogenous FVIII activity, as documented in historical medical records from a clinical laboratory demonstrating <1% FVIII coagulant activitiy or a documented genotype known to produce severe haemophilia A.
* Previous treatment for haemophilia A with any marketed recombinant and/or plasma derived FVIII for at least 150 exposure days.
* Currently receiving treatment with damoctocog alfa pegol or turoctocog alfa pegol at Screening.

Exclusion Criteria:

* Any history of a positive inhibitor test, defined as >0.6 Bethesda units (BU)/mL in at least two consecutive Bethesda inhibitor assays, or any value greated than or equal to the lower sensitivity cut-off for laboratories with cut-offs for inhibitor detection between 0.7 and 1.0 BU/mL. Family history of inhibitors will not exclude the participant.
* Positive FVIII inhibitor result (assessed by central laboratory), defined as ≥0.6 BU/mL at Screening.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Half-life (t½) of efanesoctocog alfa, damactocog alfa pegol and turoctocog alfa pegol after a single i.v. injection | up to 7 days and 14 days after the administration of the respective drugs.
  PK assessments will be based on FVIII activity levels determined by one-stage clotting assay

SECONDARY OUTCOMES:
To compare the area under the curve zero to infinity (AUC∞) of efanesoctocog alfa with that of damoctocog alfa pegol and with that of turoctocog alfa pegol after a single i.v. injection. | up to 7 days and 14 days after the administration of the respective drugs.
  The area under the curve will be calculated based on drug concentration analyses from time zero to last quantifiable sample collection timepoint
To characterize Cmax of efanesoctocog alfa and damoctocog alfa pegol or turoctocog alfa pegol after a single IV injection. | up to 7 days and 14 days after the administration of the respective drugs.
  Maximum concentration observed (Cmax) assessed by FVIII activity measurement by one-stage aPTT clotting assay
To characterize clearance of efanesoctocog alfa and damoctocog alfa pegol or turoctocog alfa pegol after a single IV injection. | up to 7 days and 14 days after the administration of the respective drugs.
  Clearance of drug/s (CL) assessed by FVIII activity measurement by one-stage aPTT clotting assay
To characterize volume of distribution of efanesoctocog alfa and damoctocog alfa pegol or turoctocog alfa pegol after a single IV injection. | up to 7 days and 14 days after the administration of the respective drugs.
  Volume of distribution (Vd) assessed by FVIII activity measurement by one-stage aPTT clotting assay
To characterize mean residence time of efanesoctocog alfa and damoctocog alfa pegol or turoctocog alfa pegol after a single IV injection. | up to 7 days and 14 days after the administration of the respective drugs.
  Mean residence time (MRT) assessed by FVIII activity measurement by one-stage aPTT clotting assay
To characterize incremental recovery of efanesoctocog alfa and damoctocog alfa pegol or turoctocog alfa pegol after a single IV injection. | up to 7 days and 14 days after the administration of the respective drugs.
  Incremental Recovery (IR) assessed by FVIII activity measurement by one-stage aPTT clotting assay
To characterize time to specific plasma FVIII levels of efanesoctocog alfa and damoctocog alfa pegol or turoctocog alfa pegol after a single IV injection. | up to 7 days and 14 days after the administration of the respective drugs.
  Time to specific plasma FVIII:C levels (40%, 20%, and 10%) assessed by FVIII activity measurement by one-stage aPTT clotting assay
To characterize time spent in plasma FVIII:C normal range for efanesoctocog alfa and damoctocog alfa pegol or turoctocog alfa pegol after a single IV injection. | up to 7 days and 14 days after the administration of the respective drugs.
  Time to spent in plasma FVIII:C normal range (50% - 150%) assessed by FVIII activity measurement by one-stage aPTT clotting assay
To evaluate the safety and tolerability of a single IV injection of efanesoctocog alfa. | From first dose of comparator to end of study, approximately 1 month.
  All safety data from visit 1 up until the dose of efanesoctocog alfa for the first treatment period and then subsequently all safety data from the dose of efanesoctocog alfa until EoS will be analyzed for this outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Santagostino, MD, Study Director — Sobi AB
Locations (7):
- Germany (2):
  - Sobi Investigational site, Frankfurt
  - Sobi Investigational Site, Oldenburg
- Italy (2):
  - Sobi Investigational Site, Milan
  - Sobi Investigational Site, Naples
- Spain (3):
  - Sobi Investigational Site, A Coruña
  - Sobi Investigational Site, Valencia
  - Sobi Investigational Site, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sobi's data sharing criteria and process for requesting access can be found at: https://www.sobi.com/en/policies
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 1 year following completion of the trial, or at the time of CSR finalization.
Access Criteria: A decision on sharing will be based on the following:
  The scientific merit of the proposal - i.e. the proposal should be scientifically sound, ethical, and have the potential to contribute to the advancement of public health.
  The feasibility of the research proposal - i.e. the requesting research team must be scientifically qualified and have the resources to conduct the proposed project.
  Maintenance of personal integrity - i.e. Sobi will not consider sharing individual data if there is a risk of re-identification of individuals despite a proper anonymisation. Moreover, the patients' informed consent will always be respected. Sobi reserves the right to reject the proposal if the anonymisation process will render unusable data.
  Publication of results - the applicants should commit to submit their findings to a peer-reviewed scientific journal, alternatively to present the results at a congress (poster or similar), regardless of the research outcome
URL: https://www.sobi.com/en/policies